CLINICAL TRIAL: NCT06793371
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of CK-4021586 in Adults With Symptomatic Heart Failure With Preserved Ejection Fraction
Brief Title: AMBER-HFpEF: Assessment of CK-4021586 in a Multi-Center, Blinded Evaluation of Safety and Tolerability Results in HFpEF
Acronym: AMBER-HFpEF
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cytokinetics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CY 9021; 2024-516349-38-00 (EU CTIS Number)
Record Dates: First submitted 2025-01-21; First posted 2025-01-27 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Symptomatic Heart Failure With Preserved Ejection Fraction (HFpEF)
Keywords: Symptomatic heart failure with preserved ejection fraction; HFpEF; Heart failure; CK-4021586; CK-586; AMBER-HFpEF; AMBER; Cardiac myosin inhibitor; CMI; CY 9021; ulacamten
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- CK-4021586 - Cohort 1 (Experimental): Participants may receive 150 mg or 300 mg of CK-4021586 daily, guided by echocardiography assessments, for 12 weeks total.
  Interventions: Drug: CK-4021586 (150 mg, 300 mg, 450 mg, and 600 mg)
- Placebo - Cohort 1 (Placebo Comparator): Participants will receive placebo daily for up to 12 weeks.
  Interventions: Drug: Placebo to match CK-4021586
- CK-4021586 - Cohort 2 (Experimental): Participants may receive 300 mg or 450 mg of CK-4021586 daily, guided by echocardiography assessments, for 12 weeks total.
  Interventions: Drug: CK-4021586 (150 mg, 300 mg, 450 mg, and 600 mg)
- Placebo - Cohort 2 (Placebo Comparator): Participants will receive placebo daily for up to 12 weeks.
  Interventions: Drug: Placebo to match CK-4021586
- CK-4021586 - Cohort 3 (Experimental): Participants may receive 450 mg or 600 mg of CK-4021586 daily, guided by echocardiography assessments, for 12 weeks total.
  Interventions: Drug: CK-4021586 (150 mg, 300 mg, 450 mg, and 600 mg)
- Placebo - Cohort 3 (Placebo Comparator): Participants will receive placebo daily for up to 12 weeks.
  Interventions: Drug: Placebo to match CK-4021586

INTERVENTIONS:
Drug: CK-4021586 (150 mg, 300 mg, 450 mg, and 600 mg) — CK-4021586 administered orally
  Other Names: ulacamten
  Arms: CK-4021586 - Cohort 1; CK-4021586 - Cohort 2; CK-4021586 - Cohort 3
Drug: Placebo to match CK-4021586 — Placebo administered orally
  Arms: Placebo - Cohort 1; Placebo - Cohort 2; Placebo - Cohort 3

SUMMARY:
This is a Phase 2 dose-finding study in adult participants with symptomatic HFpEF.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 40 years and ≤ 85 years of age at screening.
* Diagnosed with HF with NYHA functional class II or III.
* Screening echocardiography with LVEF ≥ 60%.
* Screening NT-proBNP ≥ 300 pg/mL for participants in sinus rhythm and ≥ 900 pg/mL for participants with comorbid atrial fibrillation or flutter.
* Body mass index < 40 kg/m2.
* Participants on beta-blockers, angiotensin-converting enzyme (ACE)/angiotensin II receptor blocker (ARB) or angiotensin receptor/neprilysin inhibitor (ARNI), must be on stable doses for more than 30 days prior to screening.
* Participants on a glucagon-like peptide-1 (GLP-1) agonist must be on a stable dose for more than 24 weeks prior to screening with no anticipated plans to change dose during this study.

Exclusion Criteria:

* History or evidence of any other clinically significant disorder, malignancy, active infection, other condition, or disease that, in the opinion of the investigator or the Medical Monitor, would pose a risk to patient safety or interfere with the study evaluation, procedures, or completion.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of early drug discontinuation | 12 weeks
  Incidence of early drug discontinuation observed during dosing of CK 4021586 in patients with HFpEF
Incidence of LVEF < 40% | 12 weeks
  Incidence of left-ventricular ejection fraction (LVEF) < 40% observed during dosing of CK-4021586 in patients with HFpEF
Incidence of AEs | 12 weeks
  Incidence of adverse events observed during dosing of CK-4021586 in patients with HFpEF

SECONDARY OUTCOMES:
Change in NT-proBNP | Baseline to Week 6 and Week 12
  Change from baseline values in NT-proBNP to Week 6 and Week 12
Plasma concentrations of CK-4021586 | 12 weeks
  Observed 2-hour post dose plasma concentration (C2hr) and minimum plasma concentration (Cmin) for CK-4021586 over the dosing interval
Concentration-response relationship of CK-4021586 on NT-proBNP change | Baseline to Week 12
  Slope of the relationship of plasma concentration of CK-4021586 to the change from baseline in the NT-proBNP
Concentration-response relationship of CK-4021586 to LVEF change | Baseline to Week 12
  Slope of the relationship of plasma concentration of CK-4021586 to the change from baseline in the LVEF
Change in LVEF | Baseline to Week 6 and Week 12
  Change from baseline in LVEF at Week 6 and Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Cytokinetics MD, Study Director — Cytokinetics
Locations (24):
- United States (24):
  - Eastern Shore Research Institute, LLC, Fairhope, Alabama
  - University of Arizona Sarver Heart Center, Tucson, Arizona
  - John L. McClellan Memorial Veterans Hospital, Little Rock, Arkansas
  - BioSolutions Clinical Research Center, Imperial, California
  - Profound Research LLC, Pasadena, California
  - University of California, San Francisco - Heart and Vascular Center, San Francisco, California
  - FOMAT - Comprehensive Cardiovascular Care, Santa Maria, California
  - Blue Coast Research Center, LLC, Vista, California
  - New Generation of Medical Research, Hialeah, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Louisiana Heart Center, Slidell, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University Center for Advanced Medicine, St Louis, Missouri
  - Morristown Medical Center, Morristown, New Jersey
  - NYU Langone Health, New York, New York
  - The Lindner Center for Research & Education at The Christ Hospital, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Texas Southwestern Medical Center, Dallas, Dallas, Texas
  - Center for Advanced Heart Failure, Houston, Texas
  - DelRicht Research, Vienna, Virginia
  - Swedish Heart & Vascular Institute, Advanced Cardiac Support Program, Seattle, Washington
  - Froedtert Hospital - Center for Advanced Care, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No